CLINICAL TRIAL: NCT03038113
Title: A Randomized, Sponsor-Open, Placebo-Controlled Study to Evaluate Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of Subcutaneous Administration of RO7062931 With Single Ascending Doses in Healthy Volunteers and Multiple Doses and Modified Regimens in Virologically Suppressed Patients With Chronic Hepatitis B Virus Infection
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of RO7062931in Healthy Volunteers and Subjects With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BP39405
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Results first posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — RO7062931; March8 protein, mouse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Single-Ascending Dose (SAD) (Experimental): Healthy volunteers will be enrolled in up to 8 cohorts with doses starting from 0.1 mg/kg and escalating sequentially after review of safety and pharmacokinetic (PK) data.
  Interventions: Drug: RO7062931; Drug: Placebo
- Part 2: Multiple Ascending Dose (Experimental): Participants with Chronic Hepatitis B will enrolled in Part 2. In Part 2a, participants will receive two monthly injections of either 3 doses equivalent to a multiple of the saturation dose or placebo in a 1:1:1:1 ratio. In Part 2b, a dose selected from Part 2a will be administered to participants randomized into 4 cohorts where they will be dosed weekly (QW) or bi-weekly (Q2W). Each of the cohorts in Part 2b will include participants receiving active drug or placebo in a 3:1 ratio. In Part 2c, NUC-suppressed CHB participants will receive either RO7062931+NUC for up to 24 weeks, or RO7062931+NUC+an immune modulator for up to 48 weeks, at a dose determined from Part 2a and 2b. Part 2c may also enroll treatment-naive immune-active CHB participants.
  Interventions: Drug: RO7062931; Drug: Placebo; Drug: Immune Modulator

INTERVENTIONS:
Drug: RO7062931 — Administered subcutaneously in Parts 1 and 2. Part 1 will be administered in single-ascending doses after 0.1 mg/kg starting dose. Subsequent doses of 0.3, 1, 2 and 4 mg/kg may be administered based upon tolerability. In Part 2a, participants will receive two monthly doses of either 0.4, 0.8, 1.2 times the saturation dose or placebo. In Part 2b, a dose selected from Part 2a will be administered to participants randomized into 4 cohorts QW or Q2W. In Part 2c, participants will receive RO7062831 QW on top of another therapy for up to 24 or 48 weeks.
Drug: Placebo — Part 1 cohorts: active drug vs placebo 4:1. Part 2a 4 parallel cohorts of 3 active drug doses and placebo in 1:1:1:1. Part 2b active drug vs placebo in 3:1 in 2 parallel cohorts.
Drug: Immune Modulator — Participants in Part 2c will receive an immune modulator subcutaneously QW for up to 48 weeks.
  Arms: Part 2: Multiple Ascending Dose

SUMMARY:
This randomized study will be conducted in two parts to evaluate the safety, tolerability, pharmacodynamics, and pharmacokinetics of subcutaneous administration of RO7062931. Part 1 will include only healthy participants and Part 2 will include only participants with chronic hepatitis B (CHB). Part 1 is an adaptive, single-ascending dose study with an adaptive dose-escalating schedule to determine the best dose to be evaluated in participants with CHB. Part 2 is an adaptive, parallel multiple-dose study comprised of three sub-parts which will be used to further refine the dose and dosing regimen, and to evaluate the safety and efficacy of RO7062931 when administered with standard-of-care (SoC) therapy.

ELIGIBILITY:
Inclusion Criteria:

FOR HEALTHY VOLUNTEERS ONLY - PART 1 -

* A Body Mass Index (BMI) between 18 to 30 kg/m2 inclusive and a body weight of at least 50 kg.
* Women should be of non-childbearing potential. A woman is considered to be of childbearing potential if she is post-menarcheal but has not reached a post-menopausal state and has not undergone surgical sterilization (removal of ovaries and/or uterus).
* Men must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures during treatment and up to 105 days after the last dose, and agree to refrain from donating sperm.
* Non-smoker (nor tobacco containing products) for at least 90 days prior to dosing on Day 1 and agree to remain as non-smoker during the study.

FOR CHB PARTICIPANTS ONLY - PARTS 2a and 2b:

* A BMI between 18 to 32 kg/m2 inclusive.
* Chronic hepatitis B (HBV) infection.
* Positive test for HBsAg for more than 6 months prior to randomization and HBsAg titer ≥ 10^3 IU/mL at screening.
* On entecavir, tenofovir, adefovir or telbivudine treatment for at least 6 months prior to randomization and will remain on stable treatment during the study.
* HBV deoxyribonucleic acid (DNA) ≤ 90 IU/mL for at least the preceding 6 months.
* Screening laboratory values (hematology, chemistry, urinalysis) obtained up to 56 days prior to first study treatment within normal ranges.
* Liver biopsy, fibroscan® or equivalent test obtained within the past 6 months demonstrating liver disease consistent with chronic HBV infection without evidence of bridging fibrosis or cirrhosis
* Women should be of non-childbearing potential. A woman is considered to be of childbearing potential if she is post-menarcheal but has not reached a post-menopausal state and has not undergone surgical sterilization (removal of ovaries and/or uterus).
* Men must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures during treatment and up to 105 days after the last dose, and agree to refrain from donating sperm.

FOR CHB PARTICIPANTS ONLY - PART 2c

* BMI between 18 to 32 kg/m2 inclusive
* CHB infection (HBsAg-positive for at least 6 months)
* For NUC-suppressed CHB participants: Must have been treated with a single NUC for at least 12 months, and have been on the same NUC therapy for at least 3 months prior to screening; HBV DNA <lower limit of quantification (LLOQ) at screening and in the 6 months prior to screening (at least one measurement must be >30 days prior to screening); alanine aminotransferase (ALT) </=2x upper limit of normal (ULN) for >6 months prior to screening and confirmed at screening; total bilirubin within normal range at screening, except for patients with Gilbert's syndrome
* For treatment-naive and immune-active participants: HBV DNA at screening >/=2x10^4 IU/mL for HBeAg positive participants, or >/=2x10^3 IU/mL for HBeAg negative participants; elevated serum ALT>2 ULN to </=5, 2 values within 6 months, at least one of which is at screening and that are at least 14 days apart; total bilirubin within normal range except for participants with Gilbert's syndrome
* Screening laboratory values (hematology, chemistry, urinalysis) obtained up to 28 days prior to first study treatment within normal ranges
* Liver biopsy, fibroscan, or equivalent test obtained within the last 6 months demonstrating liver disease consistent with chronic HBV infection without evidence of bridging fibrosis or cirrhosis
* Women should be of non-childbearing potential
* Men must agree to remain abstinent or use contraception, and agree to refrain from donating sperm

Exclusion Criteria:

FOR HEALTHY VOLUNTEERS ONLY - PART 1:

* History of drug or alcohol abuse or dependence in previous 6 months.
* Positive urine drug and alcohol screen or positive cotinine test at screening or Day -1.
* Positive result on hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV) 1 and 2.
* Confirmed blood pressure or resting pulse rate outside of accepted ranges.
* Participation in an investigational drug or device study within 90 days prior to screening.
* Donation of blood over 500 mL within three months prior to screening.
* Any major illness within the one month, or any febrile illness within two weeks preceding the screening visit.
* Alcohol consumption of more than 2 standard drinks per day on average.

FOR CHB PARTICIPANTS ONLY - PARTS 2a and 2b:

* History or other evidence of bleeding from esophageal varices.
* Decompensated liver disease.
* History of or suspicion of hepatocellular carcinoma or alpha fetoprotein (AFP) ≥ 13 ng/mL at Screening
* History or other evidence of a medical condition associated with chronic liver disease other than HBV infection.
* Documented history or other evidence of metabolic liver disease within one year of randomization or documented history of infection with hepatitis D virus.
* Positive test for hepatitis A (IgM anti-HAV), hepatitis C, or HIV.
* Organ transplantation.
* Significant acute infection or any other clinically significant illness within 2 weeks of randomization.
* Abnormal renal function.
* Participation in an investigational drug or device study within 30 days prior to randomization.
* Donation or loss of blood over 500 mL within 3 months prior to starting study medication.
* Administration of any blood product within 3 months of randomization.
* History or evidence of alcohol abuse (consumption of more than 2 standard drinks per day on average).

FOR CHB PARTICIPANTS ONLY - PART 2c

* History or other evidence of bleeding from esophageal varices
* Evidence of liver cirrhosis or decompensated liver disease
* One or more of the following laboratory abnormalities at screening: Total serum bilirubin > ULN (except for participants with Gilbert's disease); international normalized ratio (INR) > 1.1 ULN; serum albumin < 3.5 g/dL; AFP >13 ng/mL; positive results for anti-mitochondrial antibodies (AMA > 1:80), anti-nuclear antibody (ANA > 1:80), anti-smooth muscle antibody (ASMA > 1:40), anti-thyroperoxidase antibodies (a-TPO), anti-thyroglobulin, or anti-platelet antibodies; thyroid stimulating hormone (TSH) outside of normal range; platelet count <100,000 cells/mm^3; hemoglobin <12 g/dL (females) or <13 g/dL (males); white blood cell count <2500 cells/mm^3; and neutrophil count <1500 cells/mm^3
* History or other evidence of a medical condition associated with chronic liver disease other than HBV infection
* History of thyroid disease poorly controlled on prescribed medications or clinically relevant abnormal thyroid function tests
* Documented history or other evidence of metabolic liver disease within one year of randomization
* Positive test for hepatitis A, hepatitis C, or HIV
* History of organ transplantation
* Participation in an investigational drug or device study within 30 days prior to screening or previous treatment with an investigational agent for HBV within 6 months prior to screening
* Significant acute infection or any other clinically significant illness within 2 weeks of randomization
* Abnormal renal function, including serum creatinine > ULN or calculated creatinine clearance < 70 mL/min
* Donation or loss of blood over 500 mL within 3 months prior to randomization
* Administration of any blood product within 3 months prior to randomization
* History of alcohol abuse and/or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Australia (2):
  - Royal Melbourne Hospital, Parkville, Victoria
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin, New Territories
- New Zealand (2):
  - Auckland Clinical Studies, Auckland
  - Middlemore Hospital, Auckland
- Singapore (2):
  - National University Hospital; Dept of Gastroenterology & Hepatology, Singapore
  - Singapore General Hospital; Gastroenterology & Hepatology, Singapore
- South Korea (5):
  - Chuncheon Sacred Heart Hospital, Gangwon-Do
  - Gangnam Severance Hospital, Seoul
  - ChungAng University Hospital, Seoul
  - University of Ulsan College of Medicine, Asan Medical Center, Digestive Disease Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation - Kaohsiung Branch, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Branch, Taoyuan
- Thailand (2):
  - Siriraj Hospital; Dept. of Medicine, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gane E, Yuen MF, Kim DJ, Chan HL, Surujbally B, Pavlovic V, Das S, Triyatni M, Kazma R, Grippo JF, Buatois S, Lemenuel-Diot A, Krippendorff BF, Mueller H, Zhang Y, Kim HJ, Leerapun A, Lim TH, Lim YS, Tanwandee T, Kim W, Cheng W, Hu TH, Wat C. Clinical Study of Single-Stranded Oligonucleotide RO7062931 in Healthy Volunteers and Patients With Chronic Hepatitis B. Hepatology. 2021 Oct;74(4):1795-1808. doi: 10.1002/hep.31920. Epub 2021 Aug 25. PMID 34037271

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 - RO7062931 0.1 mg/kg: Participants received a single subcutaneous (SC) injection of 0.1 mg/kg RO7062931.
- Part 1 - RO7062931 0.3 mg/kg: Participants received a single SC injection of 0.3 mg/kg RO7062931.
- Part 1 - RO7062931 1.0 mg/kg: Participants received a single SC injection of 1.0 mg/kg RO7062931.
- Part 1 - RO7062931 2.0 mg/kg: Participants received a single SC injection of 2.0 mg/kg RO7062931.
- Part 1 - RO7062931 3.0 mg/kg: Participants received a single SC injection of 3.0 mg/kg RO7062931.
- Part 1 - RO7062931 4.0 mg/kg: Participants received a single SC injection of 4.0 mg/kg RO7062931.
- Part 1 - Placebo: Participants received a single SC injection of placebo matched to RO7062931.
- Part 2a - RO7062931 0.5 mg/kg Q1M: Participants received two QM SC injections of 0.5 mg/kg RO7062931.
- Part 2a - RO7062931 1.5 mg/kg Q1M: Participants received 2 QM SC injections of 1.5 mg/kg RO7062931.
- Part 2a - RO7062931 3.0 mg/kg Q1M: Participants received 2 QM SC injections of 3.0 mg/kg RO7062931.
- Part 2b - RO7062931 3.0 mg/kg QW: Participants received five QW SC injections of 3.0 mg/kg RO7062931.
- Part 2b - RO7062931 3.0 mg/kg Q2W: Participants received three Q2W SC injections of 3.0 mg/kg RO7062931.
- Part 2b - RO7062931 4.0 mg/kg QW: Participants received four QW SC injections of 4.0 mg/kg RO7062931.
- Part 2 - Placebo: Participants received SC placebo matched to RO7062931 over a 4-week period.
Period: Overall Study
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - Placebo | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo
Started | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 6 | 7 | 6 | 14 | 7 | 4 | 15
Completed | 8 | 8 | 7 | 8 | 8 | 8 | 11 | 6 | 7 | 6 | 14 | 7 | 4 | 14
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - Placebo | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 6 | 7 | 6 | 14 | 7 | 4 | 15 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.8 (11.9) | 29.0 (11.4) | 34.0 (11.4) | 30.4 (13.6) | 24.8 (7.9) | 23.4 (3.5) | 31.6 (9.0) | 42.0 (5.3) | 42.7 (11.1) | 47.8 (7.2) | 46.1 (12.1) | 44.9 (8.7) | 48.5 (6.9) | 44.7 (9.0) | 37.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 1 | 8
  Male | 8 | 8 | 7 | 8 | 8 | 8 | 12 | 6 | 6 | 4 | 12 | 7 | 3 | 14 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Not Hispanic or Latino | 6 | 8 | 8 | 8 | 8 | 7 | 10 | 6 | 7 | 6 | 14 | 7 | 4 | 15 | 114
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 2 | 3 | 4 | 3 | 5 | 6 | 4 | 14 | 6 | 3 | 15 | 68
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 7
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 4 | 5 | 6 | 5 | 4 | 4 | 9 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 38
  More than one race | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and AEs of Special Interest
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
  AEs of Special Interest were defined as: i.) elevated ALT/AST in combination with elevated bilirubin/clinical jaundice, ii.) suspected transmission of infectious agent by the study drug, iii.) severe injection site reactions, iv.) ALT elevation ≥10x ULN, v.) creatinine elevation ≥1.5x ULN or ≥50% from baseline.
Time Frame: Up to day 113
Population: Safety population: All study subjects that received at least one dose of study medication, whether prematurely withdrawn from the study or not.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - Placebo | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 6 | 7 | 6 | 14 | 7 | 4 | 15
Percentage of Participants
  AEs | 75.0 | 87.5 | 37.5 | 75.0 | 87.5 | 50.0 | 58.3 | 33.3 | 85.7 | 66.7 | 71.4 | 57.1 | 75.0 | 53.3
  AEs of Special Interest | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Laboratory Abnormalities Based on Hematology, Blood Chemistry, Coagulation, and Urinalysis Test Results - Part 1
Description: Marked reference range has been predefined for each laboratory parameter. The marked reference range is broader than the standard reference range. Values falling outside the marked reference range that also represent a defined change from baseline will be considered marked laboratory abnormalities (i.e., potentially clinically relevant). If a baseline value is not available for a study subject, the midpoint of the standard reference range will be used as the study participant baseline value for the purposes of determining marked laboratory abnormalities.
Time Frame: Screening, Days -1, 2, 8, 15, 29, 85
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 12
Percentage of Participants
  SGOT/AST - High | 0 | 0 | 12.5 | 0 | 0 | 0 | 0
  Chloride - Low | 0 | 0 | 0 | 0 | 0 | 0 | 8.3
  HDL Cholesterol - Low | 0 | 12.5 | 0 | 0 | 0 | 0 | 0
  Triglycerides - High | 12.5 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Laboratory Abnormalities Based on Hematology, Blood Chemistry, Coagulation, and Urinalysis Test Results - Part 2
Description: as for outcome 2
Time Frame: Screening, Days -1, 2, 8, 15, 29, at discontinuation, Days 36, 43, 57, 85, 113
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4 | 15
Percentage of Participants
  SGPT/ALT - High | 0 | 0 | 0 | 14.3 | 0 | 0 | 0
  SGOT/AST - High | 0 | 0 | 0 | 7.1 | 0 | 0 | 0
  Bicorbonate HCO3 - Low | 0 | 0 | 0 | 7.1 | 0 | 0 | 0
  Glucose, Fasting - High | 0 | 0 | 0 | 7.1 | 0 | 0 | 0
  Activated Partial Thromboplastin Time - High | 0 | 0 | 0 | 7.1 | 0 | 0 | 0
  Triglycerides - High: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Triglycerides - High | 100 |  |  |  | 0 |  |

4. Primary Outcome: Percentage of Participants With Electrocardiogram (ECG) Abnormalities Based on ECG Interpretation - Part 1
Description: Participants were monitored for clinically-significant RO7062931-related ECG changes, defined as QTcF > 500 msec, or > 60 msec longer than the pre-dose baseline, within the first 48 hours post-dose.
Time Frame: Day 1 (1,4,8,12h), Days 2 and 8, Follow Up Days 15, 29, 85
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Groups:
- Part 1 - RO7062931 0.1 mg/kg: Participants received a single SC injection of 0.1 mg/kg RO7062931.
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 12
Percentage of Participants
  Baseline | 12.5 | 50.0 | 0 | 0 | 37.5 | 25.0 | 16.7
  Day 1 - 1h | 37.5 | 50.0 | 12.5 | 25.0 | 37.5 | 25.0 | 41.7
  Day 1 - 4h | 25.0 | 25.0 | 12.5 | 25.0 | 25.0 | 12.5 | 50.0
  Day 1 - 8h | 37.5 | 50.0 | 25.0 | 12.5 | 25.0 | 25.0 | 58.3
  Day 1 - 12h | 25.0 | 50.0 | 25.0 | 25.0 | 37.5 | 12.5 | 58.3
  Day 2 - 24h | 37.5 | 50.0 | 12.5 | 12.5 | 25.0 | 25.0 | 50.0
  Day 8 - 168h | 12.5 | 50.0 | 25.0 | 37.5 | 25.0 | 25.0 | 41.7
  Follow-up Day 15 | 12.5 | 12.5 | 12.5 | 25.0 | 12.5 | 12.5 | 16.7
  Follow-up Day 29: number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 11
  Follow-up Day 29 | 25.0 | 25.0 | 14.3 | 0 | 25.0 | 25.0 | 36.4
  Extended Follow-Up: number analyzed (Participants) | 6 | 8 | 7 | 8 | 8 | 8 | 10
  Extended Follow-Up | 0 | 12.5 | 28.6 | 0 | 25.0 | 25.0 | 50.0

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) After Single Ascending Doses - Part 1
Description: Cmax values are the the peak plasma concentration reached after administration of RO7062931.
Time Frame: Days 1-8
Population: The PK analysis population included participants that did not significantly violate eligibility criteria and/or deviate significantly from the protocol. Participants with incomplete or unavailable data were excluded from analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Part 1 - RO7062931 3.0 mg/kg: Participants received a single subcutaneous (SC) injection of 3.0 mg/kg RO7062931.
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
nmol/L | 7.78 (40.2) | 19.53 (28.1) | 41.69 (30.8) | 103.68 (34.0) | 312.53 (22.2) | 153.53 (25.3)

6. Secondary Outcome: Cmax After Multiple Ascending Doses - Part 2
Description: Cmax values are the the peak plasma concentration reached after administration of RO7062931.
Time Frame: Days 1-113
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/kg
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4
mg/kg
  First Dose | 21.17 (46.4) | 72.44 (57.8) | 169.56 (43.9) | 158.61 (37.9) | 218.05 (64.4) | 232.54 (10.6)
  Last Dose | 18.56 (69.1) | 82.11 (37.6) | 194.72 (15.8) | 164.83 (65.0) | 190.83 (35.6) | 250.72 (23.4)

7. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) After Single-Ascending Doses - Part 1
Description: Tmax values are the amount of time to maximum concentration in plasma after administration of RO7062931.
Time Frame: Days 1-8
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Hours (h) | 1.75 [1.00 to 3.00] | 2.00 [1.50 to 2.00] | 3.00 [1.50 to 6.00] | 2.00 [2.00 to 6.00] | 3.00 [2.00 to 6.00] | 2.00 [2.00 to 6.00]

8. Secondary Outcome: Tmax After Multiple Ascending Doses - Part 2
Description: Tmax values are the amount of time to maximum concentration in plasma after administration of RO7062931.
Time Frame: Days 1-113
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4
Hours (h)
  First Dose | 2.98 [0.50 to 7.90] | 2.00 [2.00 to 4.00] | 2.00 [1.90 to 8.00] | 4.00 [1.90 to 6.00] | 3.98 [1.90 to 5.90] | 2.00 [1.90 to 2.00]
  Last Dose | 3.04 [2.00 to 7.70] | 3.00 [2.00 to 6.00] | 4.00 [2.00 to 4.10] | 1.97 [1.90 to 7.80] | 2.94 [1.90 to 5.70] | 2.95 [2.00 to 4.00]

9. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) After Single-Ascending Doses - Part 1
Description: AUC0-inf was calculated based on non-compartmental analysis.
Time Frame: Days 1-8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
h*nmol/L | 39.21 (14.0) | 92.72 (14.1) | 308.48 (13.2) | 792.36 (19.1) | 2478.56 (8.7) | 1257.23 (19.4)

10. Secondary Outcome: AUC0-inf After Multiple Ascending Doses - Part 2
Description: AUC0-inf was calculated based on non-compartmental analysis.
Time Frame: Days 1,22,29
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4
h*nmol/L
  Day 1: number analyzed (Participants) | 3 | 4 | 6 | 5 | 6 | 4
  Day 1 | 175.30 (6.9) | 567.07 (41.5) | 1606.49 (26.4) | 1434.39 (13.6) | 1857.98 (41.2) | 2371.66 (15.2)
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3
  Day 22 |  |  |  |  |  | 2199.57 (16.7)
  Day 29: number analyzed (Participants) | 4 | 2 | 6 | 14 | 7 | 0
  Day 29 | 180.34 (13.3) | 680.80 (8.8) | 1636.76 (11.0) | 1475.19 (30.3) | 1541.85 (26.9) |

11. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Until the Last Quantifiable Time-Point (AUC0-last) After Single Ascending Doses - Part 1
Description: AUC0-last was calculated based on non-compartmental analysis.
Time Frame: Days 1-8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (hr*nmol/L)
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 7 | 8
(hr*nmol/L) | 39.10 (14.0) | 92.62 (14.1) | 310.69 (12.9) | 789.27 (19.1) | 2448.99 (8.1) | 1253.26 (19.3)

12. Secondary Outcome: AUC0-last After Multiple Ascending Doses - Part 2
Description: AUC0-last was calculated based on non-compartmental analysis.
Time Frame: Days 1,22,29
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/L
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4
hr*nmol/L
  Day 1: number analyzed (Participants) | 6 | 7 | 6 | 6 | 7 | 4
  Day 1 | 147.30 (28.8) | 555.16 (34.8) | 1603.81 (26.4) | 1458.57 (12.9) | 1929.56 (49.9) | 2279.78 (14.7)
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4
  Day 22 |  |  |  |  |  | 2195.18 (16.6)
  Day 29: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0
  Day 29 | 141.35 (52.6) | 662.95 (20.5) | 1633.64 (11.0) | 1470.64 (30.5) | 1539.73 (27.0) |

13. Secondary Outcome: Terminal Elimination Half-Life (t1/2) After Single Ascending Doses - Part 1
Description: T1/2 was calculated based on non-compartmental analysis.
Time Frame: Days 1-8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Groups:
- Part 1 - RO7062931 3.0 mg/kg: Participants received a single subcutaneous (SC) injection of 0.1 mg/kg RO7062931.
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Hours (h) | 3.77 (65.4) | 3.99 (38.3) | 44.32 (170.4) | 97.06 (35.9) | 115.24 (60.4) | 85.70 (29.7)

14. Secondary Outcome: Terminal Elimination Half-Life (t1/2) After Multiple Ascending Doses - Part 2
Description: T1/2 was calculated based on non-compartmental analysis.
Time Frame: Days 1-113
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4
Hours (h)
  First Dose | 2.99 (13.1) | 18.81 (32.0) | 88.59 (94.1) | NA (NA) — Insufficient data to estimate parameter. | 37.96 (62.1) | 15.09 (4.3)
  Last Dose | 3.86 (107.8) | NA (NA) — Insufficient data to estimate parameter. | 119.45 (58.8) | 172.20 (26.7) | 62.08 (91.8) | 152.79 (28.7)

15. Secondary Outcome: Total Clearance (CL) After Single Ascending Doses - Part 1
Description: Apparent oral clearance was calculated from Dose/AUCinf.
Time Frame: Days 1-8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
L/h | 26.68 (21.3) | 35.97 (24.7) | 37.36 (29.9) | 26.9 (20.8) | 16.15 (18.4) | 23.46 (19.3)

16. Secondary Outcome: Total Clearance (CL) After Multiple Ascending Doses - Part 2
Description: Apparent oral clearance was calculated from Dose/AUCinf.
Time Frame: Days 1-113
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4
L/h | 31.12 (10.2) | NA (NA) — Insufficient data to estimate parameter. | 18.12 (27.2) | 21.76 (42.0) | 19.37 (43.5) | 18.75 (34.5)

17. Secondary Outcome: Volume of Distribution (Vss) After Single Ascending Doses - Part 1
Description: Vss was calculated from dose/AUCinf
Time Frame: Days 1-8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Groups:
- Part 1 - RO7062931 0.1 mg/kg: Participants received a single subcutaneous (SC) injection of 2.0 mg/kg RO7062931.
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Liters (L) | 145.22 (61.2) | 206.96 (35.2) | 2389.08 (228.8) | 3767.16 (34.4) | 2684.87 (56.8) | 2900.19 (13.9)

18. Secondary Outcome: Volume of Distribution (Vss) After Multiple Ascending Doses - Part 2
Description: Vss was calculated from dose/AUCinf
Time Frame: Days 1-113
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4
Liters (L) | 173.27 (119.8) | NA (NA) — Insufficient data to estimate parameter. | 3122.3 (46.8) | 5405.97 (53.8) | 1734.46 (86.9) | 4131.91 (22.9)

19. Secondary Outcome: Cumulative Amount Excreted Unchanged in Urine (Ae) After Single Ascending Doses - Part 1
Description: Ae: cumulative amount of drug excreted in urine over a 24 hour period or over defined time periods linked to the pools of urine collected.
Time Frame: Hours 0-4, 0-8, 0-12, and 0-24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8
pmol
  Accumulation Interval 0-4 (h) | 6180.14 (85.0) | 17111.86 (29.4) | 50248.03 (97.0) | 108870.36 (95.4) | 317169.45 (62.1) | 206781.39 (34.4)
  Accumulation Interval 0-8 (h) | 9028.41 (50.4) | 25608.73 (25.2) | 117472.78 (52.5) | 202181.27 (80.6) | 930967.60 (42.2) | 458520.65 (21.2)
  Accumulation Interval 0-12 (h) | 10399.04 (40.7) | 28335.16 (27.6) | 143182.68 (42.8) | 249381.19 (72.6) | 1148178.69 (38.2) | 592833.26 (13.5)
  Accumulation Interval 0-24 (h) | 11043.57 (38.9) | 29221.86 (28.6) | 155256.07 (38.9) | 275688.93 (68.3) | 1235241.74 (33.9) | 647368.11 (12.1)

20. Secondary Outcome: Cumulative Amount Excreted Unchanged in Urine (Ae) After Multiple Ascending Doses - Part 2
Description: as for outcome 19
Time Frame: Days 1-113
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 4.0 mg/kg QW
Number analyzed (Participants) | 6 | 7 | 6 | 7 | 14 | 4
nmol | 48.45 (22.48) | 183.38 (67.53) | 587.05 (294.65) | 790.51 (402.06) | 615.33 (432.78) | 1146.02 (177.61)

21. Secondary Outcome: Change From Baseline of Quantitative HBsAg (qHBsAg) (log10) After Multiple Ascending Doses - Part 2
Description: HBsAg is a viral parameter that can be affected by the action of RO7062931. A change from baseline in qHBsAg can indicate the drug's effect.
Time Frame: Days 1-113
Population: Participants that did not complete planned treatment and/or discontinued from the study were not included in this end point.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4 | 15
IU/mL
  Baseline value: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 4 | 13
  Baseline value | 3.39 (0.360) | 3.37 (0.272) | 3.37 (0.134) | 3.68 (0.381) | 3.76 (0.285) | 3.69 (0.274) | 3.55 (0.421)
  Final change from baseline: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 4 | 12
  Final change from baseline | -0.04 (0.057) | -0.05 (0.072) | -0.03 (0.053) | -0.09 (0.090) | -0.02 (0.070) | -0.16 (0.088) | -0.01 (0.046)

22. Secondary Outcome: Summary of Maximum qHBsAg Decrease on Days 1-113 - Part 2
Description: as for outcome 21
Time Frame: Day 1 - Day 113
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 4 | 13
IU/mL | -0.105 (0.0325) | -0.360 (0.3752) | -0.279 (0.0988) | -0.495 (0.2093) | -0.394 (0.1586) | -0.336 (0.1685) | -0.101 (0.0714)

23. Secondary Outcome: Summary of Time to Maximum qHBsAg Decrease on Day 1-113 - Part 2
Description: as for outcome 21
Time Frame: Day 1 - Day 113
Population: as for outcome 21
Measure: Median (Full Range); unit: Days
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4
Days | 49.5 [35 to 113] | 43.0 [36 to 43] | 43.0 [36 to 85] | 43.0 [29 to 113] | 39.5 [36 to 85] | 61.0 [29 to 79]

24. Primary Outcome: Percentage of Participants With Electrocardiogram (ECG) Abnormalities Based on ECG Interpretation - Part 2
Description: as for outcome 4
Time Frame: Day 1 (1,4,8h), Days 2,8,15,22 (1h and 8h), Day 23, Day 29 (1,4,8h), Day 30, Follow Up Days 36, 43, 50, 57, 78, 85, 106, 113
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4 | 15
Percentage of Participants
  Baseline | 33.3 | 14.3 | 50.0 | 50.0 | 100 | 50.0 | 46.7
  Day 1 - 1h | 66.7 | 42.9 | 50.0 | 57.1 | 85.7 | 75.0 | 40.0
  Day 1 - 4h | 33.3 | 42.9 | 66.7 | 64.3 | 57.1 | 50.0 | 33.3
  Day 1 - 8h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 7 | 4 | 15
  Day 1 - 8h | 50.0 | 0 | 33.3 | 50.0 | 100 | 25.0 | 26.7
  Day 2 - 24h | 33.3 | 28.6 | 50.0 | 57.1 | 57.1 | 50.0 | 33.3
  Day 8: number analyzed (Participants) | 6 | 7 | 6 | 14 | 6 | 4 | 15
  Day 8 | 66.7 | 57.1 | 50.0 | 57.1 | 66.7 | 25.0 | 33.3
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 14 | 6 | 4 | 7
  Day 15 |  |  |  | 50.0 | 83.3 | 50.0 | 71.4
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0 | 4 | 5
  Day 22 |  |  |  | 50.0 |  | 75.0 | 80.0
  Day 22 - 1h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Day 22 - 1h |  |  |  |  |  | 75.0 | 0
  Day 22 - 8h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Day 22 - 8h |  |  |  |  |  | 50.0 | 0
  Day 23 - 24h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Day 23 - 24h |  |  |  |  |  | 50.0 | 0
  Day 29: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 | 66.7 | 50.0 | 83.3 | 50.0 | 83.3 |  | 50.0
  Day 29 - 1h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 - 1h | 83.3 | 16.7 | 50.0 | 64.3 | 83.3 |  | 58.3
  Day 29 - 4h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 - 4h | 50.0 | 33.3 | 16.7 | 57.1 | 66.7 |  | 25.0
  Day 29 - 8h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 - 8h | 16.7 | 0 | 66.7 | 64.3 | 66.7 |  | 16.7
  Day 30 - 24h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 30 - 24h | 66.7 | 16.7 | 100 | 50.0 | 66.7 |  | 41.7
  Follow-up Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 36 |  |  |  |  |  | 75.0 | 0
  Follow-up Day 43: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 13
  Follow-up Day 43 | 83.3 | 14.3 | 16.7 | 57.1 | 57.1 |  | 38.5
  Follow-up Day 50: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 50 |  |  |  |  |  | 50.0 | 0
  Follow-up Day 57: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 13
  Follow-up Day 57 | 66.7 | 14.3 | 66.7 | 57.1 | 71.4 |  | 53.8
  Follow-up Day 78: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 78 |  |  |  |  |  | 25.0 | 0
  Follow-up Day 85: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Follow-up Day 85 | 33.3 | 14.3 | 66.7 | 50.0 | 57.1 |  | 38.5
  Follow-up Day 106: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 106 |  |  |  |  |  | 50.0 | 0
  Follow-up Day 113: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Follow-up Day 113 | 66.7 | 14.3 | 50.0 | 42.9 | 71.4 |  | 46.2

25. Primary Outcome: Percentage of Participants With T-Wave Abnormalities Based on T-Wave Assessment - Part 1
Description: Table entries provide the percentage of participants with abnormalities during treatment assessment. Abnormalities reported in participants with missing baseline values are included. Baseline is the Participant's last observation prior to initiation of study drug.
Time Frame: Day 1 (1,4,8,12h), Days 2 and 8, Follow Up Days 15, 29, 85
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 12
Percentage of Participants
  Baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 - 1h | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 - 4h | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 - 8h | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 - 12h | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 2 - 24h | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 - 168h | 0 | 0 | 0 | 0 | 12.5 | 0 | 0
  Follow-up Day 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-up Day 29: number analyzed (Participants) | 8 | 8 | 7 | 8 | 8 | 8 | 11
  Follow-up Day 29 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Extended Follow-Up: number analyzed (Participants) | 6 | 8 | 7 | 8 | 8 | 8 | 10
  Extended Follow-Up | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Primary Outcome: Percentage of Participants With U-Wave Abnormalities Based on U-Wave Assessment - Part 1
Description: as for outcome 25
Time Frame: Day 1 (1,4,8,12h), Days 2 and 8, Follow Up Days 15, 29, 85
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 12
Percentage of Participants
  Baseline | 12.5 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 - 1h | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 - 4h | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 - 8h | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 - 12h | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 2 - 24h | 12.5 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 - 168h | 0 | 0 | 0 | 0 | 12.5 | 0 | 0
  Follow-up Day 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-up Day 29: number analyzed (Participants) | 8 | 8 | 7 | 8 | 8 | 8 | 11
  Follow-up Day 29 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Extended Follow-Up: number analyzed (Participants) | 6 | 8 | 7 | 8 | 8 | 8 | 10
  Extended Follow-Up | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Primary Outcome: Percentage of Participants With T-Wave Abnormalities Based on T-Wave Assessment - Part 2
Description: as for outcome 25
Time Frame: as for outcome 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4 | 15
Percentage of Participants
  Baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 - 1h | 0 | 0 | 16.7 | 0 | 0 | 0 | 0
  Day 1 - 4h | 0 | 0 | 33.3 | 7.1 | 0 | 0 | 0
  Day 1 - 8h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 7 | 4 | 15
  Day 1 - 8h | 0 | 0 | 16.7 | 0 | 0 | 0 | 0
  Day 2 - 24h | 0 | 0 | 16.7 | 0 | 0 | 0 | 0
  Day 8: number analyzed (Participants) | 6 | 7 | 6 | 14 | 6 | 4 | 15
  Day 8 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 14 | 6 | 4 | 7
  Day 15 |  |  |  | 7.1 | 0 | 0 | 0
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0 | 4 | 5
  Day 22 |  |  |  | 7.1 |  | 0 | 0
  Day 22 - 1h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Day 22 - 1h |  |  |  |  |  | 0 | 0
  Day 22 - 8h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Day 22 - 8h |  |  |  |  |  | 0 | 0
  Day 23 - 24h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Day 23 - 24h |  |  |  |  |  | 0 | 0
  Day 29: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 | 0 | 0 | 16.7 | 0 | 0 |  | 0
  Day 29 - 1h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 - 1h | 0 | 0 | 16.7 | 0 | 0 |  | 8.3
  Day 29 - 4h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 - 4h | 0 | 0 | 0 | 7.1 | 0 |  | 8.3
  Day 29 - 8h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 - 8h | 0 | 0 | 16.7 | 0 | 0 |  | 0
  Day 30 - 24h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 30 - 24h | 0 | 0 | 16.7 | 0 | 0 |  | 0
  Follow-up Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 36 |  |  |  |  |  | 0 | 0
  Follow-up Day 43: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 13
  Follow-up Day 43 | 0 | 0 | 16.7 | 7.1 | 0 |  | 0
  Follow-up Day 50: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 50 |  |  |  |  |  | 0 | 0
  Follow-up Day 57: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 13
  Follow-up Day 57 | 0 | 0 | 16.7 | 7.1 | 0 |  | 0
  Follow-up Day 78: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 78 |  |  |  |  |  | 0 | 0
  Follow-up Day 85: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 13
  Follow-up Day 85 | 0 | 0 | 16.7 | 0 | 0 |  | 0
  Follow-up Day 106: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 106 |  |  |  |  |  | 0 | 0
  Follow-up Day 113: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 13
  Follow-up Day 113 | 0 | 0 | 0 | 0 | 0 |  | 0

28. Primary Outcome: Percentage of Participants With U-Wave Based on U-Wave Assessment - Part 2
Description: as for outcome 25
Time Frame: as for outcome 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4 | 15
Percentage of Participants
  Baseline | 0 | 14.3 | 0 | 7.1 | 0 | 25.0 | 6.7
  Day 1 - 1h | 0 | 14.3 | 0 | 7.1 | 0 | 25.0 | 6.7
  Day 1 - 4h | 16.7 | 14.3 | 0 | 7.1 | 0 | 25.0 | 6.7
  Day 1 - 8h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 7 | 4 | 15
  Day 1 - 8h | 0 | 16.7 | 0 | 7.1 | 0 | 25.0 | 6.7
  Day 2 - 24h | 0 | 14.3 | 0 | 7.1 | 0 | 25.0 | 6.7
  Day 8: number analyzed (Participants) | 6 | 7 | 6 | 14 | 6 | 4 | 15
  Day 8 | 16.7 | 14.3 | 0 | 7.1 | 0 | 25.0 | 6.7
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 14 | 6 | 4 | 7
  Day 15 |  |  |  | 7.1 | 0 | 25.0 | 0
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0 | 4 | 5
  Day 22 |  |  |  | 7.1 |  | 25.0 | 0
  Day 22 - 1h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Day 22 - 1h |  |  |  |  |  | 25.0 | 0
  Day 22 - 8h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Day 22 - 8h |  |  |  |  |  | 25.0 | 0
  Day 23 - 24h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Day 23 - 24h |  |  |  |  |  | 25.0 | 0
  Day 29: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 | 0 | 16.7 | 0 | 7.1 | 0 |  | 0
  Day 29 - 1h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 - 1h | 0 | 16.7 | 0 | 7.1 | 0 |  | 0
  Day 29 - 4h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 - 4h | 0 | 16.7 | 0 | 7.1 | 0 |  | 0
  Day 29 - 8h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 29 - 8h | 0 | 16.7 | 0 | 7.1 | 0 |  | 0
  Day 30 - 24h: number analyzed (Participants) | 6 | 6 | 6 | 14 | 6 | 0 | 12
  Day 30 - 24h | 0 | 16.7 | 0 | 7.1 | 0 |  | 0
  Follow-up Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 36 |  |  |  |  |  | 25.0 | 0
  Follow-up Day 43: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 13
  Follow-up Day 43 | 0 | 0 | 0 | 7.1 | 0 |  | 0
  Follow-up Day 50: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 50 |  |  |  |  |  | 25.0 | 0
  Follow-up Day 57: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 13
  Follow-up Day 57 | 0 | 14.3 | 0 | 7.1 | 0 |  | 7.1
  Follow-up Day 78: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 78 |  |  |  |  |  | 25.0 | 0
  Follow-up Day 85: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 13
  Follow-up Day 85 | 0 | 14.3 | 0 | 7.1 | 0 |  | 7.1
  Follow-up Day 106: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Follow-up Day 106 |  |  |  |  |  | 25.0 | 0
  Follow-up Day 113: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 13
  Follow-up Day 113 | 0 | 14.3 | 0 | 7.1 | 14.3 |  | 15.4

29. Primary Outcome: Percentage of Participants With QTcF Values Between 450 Msec - 480 Msec - Part 2
Description: as for outcome 25
Time Frame: as for outcome 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 4 | 15
Percentage of Participants
  Baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 - 1h | 0 | 0 | 0 | 0 | 14.3 | 0 | 0
  Day 1 - 4h | 0 | 0 | 0 | 0 | 14.3 | 0 | 0
  Day 1 - 8h | 0 | 0 | 0 | 0 | 14.3 | 0 | 0
  Day 2 - 24h | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 | 0 | 0 | 0 | 7.1 | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 14 | 7 | 4 | 15
  Day 15 |  |  |  | 0 | 0 | 0 | 0
  Day 22: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0 | 4 | 15
  Day 22 |  |  |  | 7.1 |  | 0 | 0
  Day 22 - 1h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 15
  Day 22 - 1h |  |  |  |  |  | 25.0 | 0
  Day 22 - 8h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 15
  Day 22 - 8h |  |  |  |  |  | 0 | 0
  Day 23 - 24h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 15
  Day 23 - 24h |  |  |  |  |  | 0 | 0
  Day 29: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Day 29 | 0 | 0 | 16.7 | 7.1 | 0 |  | 8.3
  Day 29 - 1h: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Day 29 - 1h | 0 | 0 | 33.3 | 7.1 | 0 |  | 8.3
  Day 29 - 4h: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Day 29 - 4h | 0 | 0 | 33.3 | 7.1 | 0 |  | 8.3
  Day 29 - 8h: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Day 29 - 8h | 0 | 0 | 0 | 7.1 | 0 |  | 0
  Day 30 - 24h: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Day 30 - 24h | 0 | 0 | 0 | 7.1 | 0 |  | 8.3
  Follow-up Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 15
  Follow-up Day 36 |  |  |  |  |  | 0 | 0
  Follow-up Day 43: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Follow-up Day 43 | 0 | 0 | 0 | 7.1 | 0 |  | 0
  Follow-up Day 50: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 15
  Follow-up Day 50 |  |  |  |  |  | 0 | 0
  Follow-up Day 57: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Follow-up Day 57 | 0 | 0 | 50.0 | 7.1 | 0 |  | 0
  Follow-up Day 78: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 15
  Follow-up Day 78 |  |  |  |  |  | 0 | 0
  Follow-up Day 85: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Follow-up Day 85 | 0 | 14.3 | 33.3 | 7.1 | 14.3 |  | 7.7
  Follow-up Day 106: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 15
  Follow-up Day 106 |  |  |  |  |  | 0 | 0
  Follow-up Day 113: number analyzed (Participants) | 6 | 7 | 6 | 14 | 7 | 0 | 15
  Follow-up Day 113 | 0 | 0 | 33.3 | 0 | 14.3 |  | 0

ADVERSE EVENTS:
Time Frame: Approximately 32 months
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and does not necessarily require a causal relationship with treatment. An adverse event can be any unfavorable and unintended sign, symptom, or disease temporally associated with use of a pharmaceutical product, whether or not considered related to the product. Preexisting conditions that worsen during a study are also considered adverse events.
Arm/Group | Part 1 - RO7062931 0.1 mg/kg | Part 1 - RO7062931 0.3 mg/kg | Part 1 - RO7062931 1.0 mg/kg | Part 1 - RO7062931 2.0 mg/kg | Part 1 - RO7062931 3.0 mg/kg | Part 1 - RO7062931 4.0 mg/kg | Part 1 - Placebo | Part 2a - RO7062931 0.5 mg/kg Q1M | Part 2a - RO7062931 1.5 mg/kg Q1M | Part 2a - RO7062931 3.0 mg/kg Q1M | Part 2b - RO7062931 3.0 mg/kg QW | Part 2b - RO7062931 3.0 mg/kg Q2W | Part 2b - RO7062931 4.0 mg/kg QW | Part 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/6 | 0/7 | 0/6 | 0/14 | 0/7 | 0/4 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/6 | 0/7 | 0/6 | 0/14 | 0/7 | 0/4 | 0/15
Other Adverse Events (participants affected / at risk) | 6/8 | 7/8 | 3/8 | 6/8 | 7/8 | 4/8 | 7/12 | 2/6 | 6/7 | 4/6 | 10/14 | 4/7 | 3/4 | 8/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - RO7062931 0.1 mg/kg (N=8) | Part 1 - RO7062931 0.3 mg/kg (N=8) | Part 1 - RO7062931 1.0 mg/kg (N=8) | Part 1 - RO7062931 2.0 mg/kg (N=8) | Part 1 - RO7062931 3.0 mg/kg (N=8) | Part 1 - RO7062931 4.0 mg/kg (N=8) | Part 1 - Placebo (N=12) | Part 2a - RO7062931 0.5 mg/kg Q1M (N=6) | Part 2a - RO7062931 1.5 mg/kg Q1M (N=7) | Part 2a - RO7062931 3.0 mg/kg Q1M (N=6) | Part 2b - RO7062931 3.0 mg/kg QW (N=14) | Part 2b - RO7062931 3.0 mg/kg Q2W (N=7) | Part 2b - RO7062931 4.0 mg/kg QW (N=4) | Part 2 - Placebo (N=15)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 4 (7) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 2 (3) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Clavicle feacture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03038113/Prot_SAP_000.pdf